CLINICAL TRIAL: NCT00813254
Title: Quality of Life and Cost Utility Analysis in the Treatment of Recurrent, Platinum-Resistant Ovarian Cancer
Brief Title: Cost Utility Analysis in Recurrent Ovarian Cancer
Status: Withdrawn | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0611
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Ovarian Cancer
Keywords: Platinum-Resistant Ovarian Cancer; Platinum-based chemotherapy; Ovarian Cancer; Ovary; Epithelial ovarian cancer; Quality of Life; Cost Utility Analysis; Sexual functioning; Questionnaire; Caregiver
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire: Longitudinal measure of QOL, sexual functioning and symptoms in women with recurrent, platinum-resistant ovarian cancer receiving multiple second-line treatment regimens
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires 1 - 5 will be completed on Day 1 of study as a Baseline.
  Other Names: Survey

SUMMARY:
The goal of this research study is to learn about the quality of life and sexual functioning of women with platinum-resistant ovarian cancer as they receive other treatments for the disease.

Researchers will study the costs for chemotherapy treatments, other medical expenses, and treatment-related expenses that are not medical. Researchers will also review any symptoms these patients may experience related to the cancer or treatment.

In addition, researchers want to learn if and how these patients' caregivers feel the status of these patients' health may have affected the caregivers' productivity at work and at home.

DETAILED DESCRIPTION:
Study Participation:

If you agree to take part in this study, medical and demographic information will be collected from your medical record and/or by asking you in person when you come to the clinic for your routine visits. This information includes your date of birth, medical history, occupation, marital status, race, household income, and number of children and/or other dependents (if any).

On Day 1 of your study participation, you will be interviewed by a research staff member. In this interview, you will be asked about your health and any symptoms related to the cancer and/or cancer treatment. You will also be asked for the best way of contacting you. This interview should take about 30 minutes to complete. After the interview, you will complete a set of 5 questionnaires. In total, the questionnaires should take about 15 minutes to complete. You will repeat these same 5 questionnaires on Day 1 of each of your chemotherapy cycles. The questionnaires include the following:

* Questionnaire 1 (The Short Form 12) asks about your physical and emotional health, any pain, social functioning, and general health. This information will help researchers keep track of how you feel and how well you are able to do your usual activities.
* Questionnaire 2 (The Functional Assessment of Cancer Therapy) asks about the symptoms of cancer and how these symptoms may affect your physical, social, and emotional well-being.
* Questionnaire 3 (Medical Outcomes Study) asks about your sexual functioning. Researchers believe this information is important in understanding how health problems affect people's lives.
* Questionnaire 4 (The Functional Assessment of Cancer Therapy/Neurotoxicity questionnaire) asks whether or not you have had any numbness and/or tingling in your hands and/or feet. This numbness/tingling can occur as a side effect of some chemotherapy drugs that are commonly given to patients with ovarian cancer.
* Questionnaire 5 (The Memorial Symptom Assessment Scale) asks about the symptoms of ovarian cancer and the side effects of ovarian cancer treatment.

In addition, you will also be asked to complete the following questionnaires for each cycle of chemotherapy:

* Questionnaire 6 (The Productivity and Activity Impairment General Health questionnaire) asks about how you feel your health status may have affected your and/or your primary caregiver's "productivity" (your ability to perform normal activities) at work and at home.
* Questionnaire 7 (The European Quality of Life instrument) asks a few questions about your health status on that particular day. It also asks you to rate your health status by marking on a scale how good or bad your health is on that day.
* Questionnaire 8 is a diary in which you will record all medical costs (such as any emergency room visits, hospitalizations, doctor's visits, and medications) that you have had to pay for in the last week.
* Questionnaire 9 is a diary in which you will record your treatment-related costs that are not medical (such as travel, child care costs, parking fees, and gasoline).

You can bring the completed Questionnaires 6-9 with you when you return for your next follow-up visit, email, fax or mail them back to the clinic before your next visit. If necessary, you may complete them over the phone instead. In total, Questionnaires 6-9 should take about 7 minutes to complete each time.

Questionnaire Content:

Your responses on these questionnaires will not be shared with the doctor who is treating you for cancer. If you feel you need a doctor's opinion about anything that is asked about in these questionnaires (such as cancer symptoms or mental or emotional difficulties), please contact your doctor.

If your questionnaire responses show that you may be having emotional difficulties or depression, you will be provided with names of mental health providers in case you would like to receive a mental health screening.

Caregivers' Participation:

Your caregiver will also be asked to complete Questionnaire 6 for each cycle of chemotherapy you receive. Specifically, the caregiver will answer questions about how he or she feels your health status may have affected his or her productivity at work and at home.

Your questionnaires will be used for research purposes only, and your responses will not be shared with the caregiver. Likewise, the caregiver's responses will not be shared with you. You will receive separate return envelopes for mailing back your questionnaires separately from the caregiver's.

Length of Study Participation:

This is a long-term study, and you will remain "on study" for as long as you and the caregiver agree to keep filling out the questionnaires. If you stop receiving treatment for the cancer, your and the caregiver's participation in this study will be over.

This is an investigational study. You will receive stamped, self-addressed envelopes for mailing the questionnaires back to the clinic.

Up to 43 patients and 43 caregivers will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent, platinum-resistant epithelial ovarian cancer who are beginning any second-line treatment
2. Patients must be English-speaking
3. Patients must be able to read and write English
4. Patients receiving all chemotherapy at MD Anderson Cancer Center

Exclusion Criteria:

1. Patients with non-epithelial ovarian cancers including sex-cord stromal tumors, germ cell tumors, low-grade tumors, and metastatic disease to the ovary
2. Patients who are receiving protocol therapy
3. Patients who have had a prior diagnosis of invasive cancer at other sites (excluding basal cell carcinoma of the skin)
4. Patients who are receiving radiation therapy as a treatment modality

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female study participants that were diagnosed with Ovarian Cancer that are now "Platinum-Resistant."
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Mean Score for the FACT-O instrument | First 2 days of chemotherapy cycles
  Participants will complete questionnaires 1 - 5 at baseline and Day 1 of each of their chemotherapy cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Frumovitz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org